CLINICAL TRIAL: NCT00303238
Title: Double-Blind Trial to Evaluate the Effect of Botanical Dietary Supplements on C-Reactive Protein, Ex-Vivo IL-1 Production, and In-Vivo IL-1 Gene Expression in Healthy Human Subjects
Brief Title: Study to Evaluate the Effect of Botanical Dietary Supplements on Inflammation in Healthy People
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Access Business Group (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: Lakeside 3a
Record Dates: First submitted 2006-03-14; First posted 2006-03-16 (Estimated); Last update posted 2006-03-16 (Estimated); Status verified 2006-03

CONDITIONS: Healthy
Keywords: Inflammation; Interleukin-1; C-reactive protein; Genotype; Rose Hips; Blueberry; Blackberry; Aframomum melegueta; Resveravine
MeSH Terms: conditions — Inflammation | interventions — blueberry extract

INTERVENTIONS:
Drug: Rose hips extract + blueberry/blackberry extract + resveravine
Drug: Rose hips extract + blueberry/blackberry extract + Aframomum melegueta extract
Drug: Rose hips extract + resveravine + Aframomum melegueta extract

SUMMARY:
The purpose of the study is to evaluate the effect of botanical dietary supplements on inflammation in healthy people with different genetic responses to inflammation.

DETAILED DESCRIPTION:
The impact of nutrition and lifestyle have long been recognized as key determinants of risk for chronic degenerative diseases such as atherosclerosis, osteoporosis, rheumatoid arthritis, etc. While it is clear that reducing nutrition and lifestyle risk factors for a particular disease reduces risk in populations, individuals differ significantly in the degree to which presumed beneficial changes in these risk factors confer risk or lack thereof. This individual response is increasingly thought to be due genetic differences.

Developing in parallel with the research on genetic impact and chronic disease risk is a strengthening body of data suggesting that inflammation is common to many chronic degenerative diseases. A key cytokine regulator of the inflammatory response, interleukin-1 (IL-1), has emerged as playing a particularly important role at the genetic level in determining the degree to which the inflammation pathway is turned on. The strong influence of IL-1 over the inflammation pathway follows from its functional role as one of the initiating cytokine signals in the inflammatory pathway. Recent research has identified polymorphisms in the IL-1 gene that lead to over expression of IL-1 and elevated levels of the inflammation biomarker, c-reactive protein (CRP). Individuals with selected polymorphisms associated with over expression of IL-1 appear to be at increased risk for selected chronic degenerative diseases.

The mechanistic role of IL-1 in the overall inflammatory response and the detrimental impact of IL-1 over-expression may create a need for IL-1 genotype-directed nutritional, lifestyle and dietary supplement interventions that address the individual genetic risk for inflammation associated diseases by reducing chronic inflammation.

The current protocol draws participants from a pre-existing database containing information on health and lifestyle, IL-1 genotype, and inflammation biomarkers from approximately 2300 people. The database was created under a separate IRB-approved protocol. Participants will randomly receive one of three botanical formulas or a placebo once a day for 20 weeks. The effects of the botanical formulas on recognized markers of inflammation, e.g., CRP, as well as surrogate readouts of the inflammation pathway, ex vivo IL-1 production, and in vivo expression of the IL-1 gene will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

1. Non-smoking adults aged 18 and up
2. Individual should be judged to be in good general health on the basis of an interview, vitals assessment, and physical examination
3. Individual is willing to maintain their normal dietary and exercise habits throughout the duration of the trial
4. Individual understands the procedures and agrees to participate in the study
5. Individual is able and willing to provide written informed consent
6. Average serum CRP level between 2 and 10 mg/L inclusively.

Exclusion Criteria:

1. Current smoker or history of tobacco use within the past year
2. Use of dietary supplements within one week of Day 1. Supplements include any vitamins, minerals, and herbal products, including herbal drinks
3. Presence of, or clinical significant history of, autoimmune, blood, cancer, cardiovascular, endocrine, kidney, liver, lung, gastrointestinal, metabolic disorder, and/or any other chronic health condition identified from the findings of the interview
4. Currently treated for uncontrolled hypertension or blood pressure > 170 mm Hg systolic or > 100 mm Hg diastolic during seated, resting measurement on two consecutive occasions during visit 1
5. Therapeutic use of nitroglycerin, alpha1- or beta-adrenergic blockers, Apresoline, Loniten, calcium channel blockers, ACE inhibitors, and/or any other drug that may alter blood pressure
6. Therapeutic use of coumadin, aspirin, or other medications that influence blood coagulation
7. Current use of NSAIDS, including COX-2 inhibitors
8. Therapeutic use of cholesterol-lowering medications such as HMG CoA reductase inhibitors, bile acid binding agents, bile acid binding resins, nicotinic acid, and fibric acid derivatives
9. Known allergy to rose hips, blueberries, blackberries, resveravine, and/or A. melegueta
10. Current use of any form of steroid drug (prescription or non-prescription), including inhalers for asthma
11. Current use of any form of hormone replacement therapy (HRT and ERT)
12. Participation in another clinical trial within 30 days of enrollment into the study
13. History or current abuse of drugs or alcohol, or intake > 2 alcoholic beverages per day
14. Pregnant or lactating women, or women of child-bearing potential unwilling to use a medically approved form of birth control
15. Any condition that the Principal Investigator believes may put the subject at undue risk
16. Serum CRP less than 3 or higher than 10 mg/L. If a subject has a CRP > 10 mg/L at screening, the measurement will be repeated two weeks later to determine whether the subject should be excluded from the protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200
Dates: Start 2004-10; Study Completion 2005-12

PRIMARY OUTCOMES:
- Serum C-reactive protein levels
- In vivo IL-1 gene expression
- Ex vivo IL-1 production

SECONDARY OUTCOMES:
- Cytokine Inflammatory Panel (IL-1-alpha, TNF-alpha, IL-6, IL-8, IL-10, and IL-12)
- Serum Amyloid A (SAA)
- Serum Intracellular Adhesion Molecule-1 (ICAM-1)
- Fibrinogen

CONTACTS AND LOCATIONS:
Overall Officials: Russell K Randolph, PhD, Study Chair — Access Business Group, LLC; Kenneth Kornman, PhD, Study Director — Interleukin Genetics
Locations (8):
- United States (8):
  - Sall Research Medical Center, Artesia, California
  - Southbay Pharma Research, Buena Park, California
  - Access Business Group, LLC, Buena Park, California
  - Providence Clinical Research, Burbank, California
  - National Institute of Clinical Research, Los Angeles, California
  - East Coast Clinical Research, Haverhill, Massachusetts
  - Alticor, Inc, Ada, Michigan
  - Omega Medical Research, Warwick, Rhode Island